CLINICAL TRIAL: NCT00312559
Title: The Therapeutic Effects of Yoga in Individuals With Parkinson's Disease
Brief Title: The Therapeutics Effects of Yoga in Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 10214
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2007-08-20 (Estimated); Status verified 2007-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Behavioral: Yoga Training

SUMMARY:
To determine if yoga is beneficial in improving physical function quality of life and medical status in people with Parkinson's disease

DETAILED DESCRIPTION:
This pilot study is a randomized controlled study of 20-30 individuals with Parkinson's disease will have a control group with no training and a research group with yoga training. The control group will have the opportunity to attend yoga training of the same intensity after the study is completed. The effects of yoga will not be on the control group. Data on physical function will be derived from assessments including strength, balance, flexibility, ROM. gait, posture and functional analysis performed in the Georgia Holland Cardiopulmonary and Neuromuscular Research Lab. Questionnaires related to quality of life, depression and falls will determine psychological impact or yoga training. Vital signs, pulmonary function tests and blood draws will be done in the General Clinical research Center (GCRC) and protein analysis will be done in the diabetes research lab.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease
* Stage 1-3 Hoehn & Yahr

Exclusion Criteria:

* Decline in immune function
* 6 month joint surgery
* spinal fusions
* decline in mental status measured by Folstein Mini Mental Status Exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2006-02; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test, serum protein levels BP, HR, RR, strength testing using microFET, flexibility and range of motion testing using goniometer, balance/posture gait optitrk system, Berg balance scale

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale
Hoehn & Yahr Classification Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Searls, PT, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States